CLINICAL TRIAL: NCT03149744
Title: A Mixed-methods Evaluation of a Novel Apnoea Event Detection Monitor in Comparison to Standard of Care Limited Overnight Polysomnography
Brief Title: Mixed Methods Evaluation of a Novel Apnoea Event Detection Monitor
Status: Completed | Type: Observational
Sponsor: PMD Solutions (Industry)
Collaborators: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: PMD-CS-008
Record Dates: First submitted 2017-05-09; First posted 2017-05-11 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Respiratory Rate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: RespiraSense Sleep Screener — RespiraSense will be worn at the same time as the standard of care SomnoScreen and it's results will be masked to the site team

SUMMARY:
This investigation is looking at a currently available technology to see if it could have another use i.e. in helping to diagnose patients with sleep apnoea.

With 2-4% of the population suffering from this disease, and the current wait time for a test at approximately 20 weeks, it is hoped that a simple screening method could help speed up the process of finding these patients and getting them on treatment faster.

The current standard of care test involves a sleep study in the patients own home with a device with multiple parts and wires. The RespiraSense Sleep Screener is completely cableless and consists of one small, discrete unit attached to the patients side and a mobile device plugged in by the bed.

Patients at Queen Alexandra Hospital who are prescribed sleep studies will be invited to participate. The RespiraSense Sleep Screener data is only for comparison purposes and will have no effect on their clinical care.

If patients agree to participate they will undergo the sleep study with both devices in the same night and may be followed up with over the phone on their experiences with the test.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 Years
* Patients due to undergo home monitoring to investigate presence of sleep apnoeic events
* Patients able to provide informed consent to participate in this investigation

Exclusion Criteria:

* Patients with known respiratory disorders that are uncontrolled at the time of the sleep study
* Patients allergic to medical grade skin adhesive
* Patients on long term, oral steroid use
* Pregnant women during second and third trimester
* Patients presently on any sleep disorder therapy
* Patients with any history of substance abuse (drug or alcohol) that may interfere with their ability to cooperate and comply with the investigation procedures
* Patients with any disorder, including cognitive dysfunction, which would affect the ability to accurately complete questionnaires and freely give full informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients due to undergo standard of care home sleep testing
Sampling Method: Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2017-02-28 (Actual); Primary Completion 2017-05-02 (Actual); Study Completion 2017-05-02 (Actual)

PRIMARY OUTCOMES:
Similarity to standard of care | One night
  The mean error of the device relative to the overnight polysomnography tests ≥ 10 AHI

SECONDARY OUTCOMES:
Qualitative evaluation of RespiraSense | One night
  to qualitatively evaluate the perceptions, values and opinions of the RS Sleep Screener device compared with the comparator to identify potential modifications to improve patient acceptance and to inform future implementation of the device within the NHS setting

CONTACTS AND LOCATIONS:
Overall Officials: Anoop Chauhan, Principal Investigator — Portsmouth Hospitals NHS Trust
Locations (1):
- Queen Alexandra Hospital, Portsmouth, United Kingdom

IPD SHARING:
Plan to Share IPD: No